CLINICAL TRIAL: NCT02925039
Title: The "Feedback Integrated Rehabilitation for Sit-to-stand Training": a Pilot Randomised Controlled Trial Testing Clinical Acceptability and Effectiveness
Brief Title: Sit-to-stand Exercise Training With Performance Feedback
Acronym: FIRST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Strathclyde (Other)
Responsible Party: Principal Investigator, Andrew Kerr, Lecturer, University of Strathclyde
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UStrathclydeBMEKerr01
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Geriatric Diseases
Keywords: Rehabilitation; Geriatric
MeSH Terms: interventions — Rehabilitation; Therapeutics

STUDY DESIGN:
Intervention Model Description: Pilot Randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Sit to stand training augmented with technology delivered movement feedback
  Interventions: Other: Rehab with computer feedback
- Control (Active Comparator): Sit to stand training as per normal practice
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Rehab with computer feedback — Sit to stand training with addition of computerised feedback (speed, symmetry and trunk tilt)
  Arms: Experimental
Other: Treatment as usual — Treatment as usual
  Arms: Control

SUMMARY:
The sit-to-stand (STS) movement is a key functional movement critical to independent living. This movement is physically demanding to conduct, especially in older adults, and in the presence of physical impairments associated with a range of conditions, such as stroke, osteoarthritis, Parkinson disease and hip arthroplasty. A limited capacity to perform this movement increases the risk of falls, dependency and increased support for personal care and rehabilitation. Restoring independence in this movement is, therefore, considered a priority for physical rehabilitation.

Sit-to-stand capacity can be regained through participating in rehabilitation exercises. Providing feedback on performance of this movement could enhance the training. Thus, it is an essential aspect of physical therapy. Healthcare providers are required to meet the needs of an increasingly frail population as well as meeting national, evidence-based, guidelines for improving outcomes in conditions such as stroke which includes an increase in the practice repetition of functional movements. Reliance on rehabilitation staff to provide practice, however, places a limit on practice volume, potentially restricting outcomes. Using technology to enhance safe, repetitive practice of this movement with minimal supervision from skilled professionals would be beneficial to patients and rehabilitation services.

The primary aim of this study is to test the acceptability and feasibility of a STS training system that enhances movement feedback to patients undergoing rehabilitation. A secondary aim is to gather data on the effectiveness of the system compared to conventional rehabilitation. This information will inform a statistically powered phase 2 trial.

DETAILED DESCRIPTION:
Research Design:

This is a pilot randomised controlled study to test the acceptability and feasibility of a sit-to-stand (STS) training system and gather preliminary data on its effectiveness. Participants will be randomly allocated to an experimental group where participants will receive sit to stand training enhanced by the feedback system or a control group where participants will receive the usual sit to stand training as provided by the treating therapist.

Participants and recruitment:

Patients with physical impairments that affect their capacity to perform the STS movement and who are about to start active rehabilitation will be identified by the clinical team on the ward. If individuals identified in this way indicate to the clinical team that they are willing to talk to the researcher about the study a mutually convenient time will be arranged for the researcher to speak individually to the patient about the study. An information sheet will be left with the patient and they will be encouraged to read this and speak to family and friends about their possible participation. No less than 48 hours after the information sheet is provided, the researcher will make contact with the patient to discuss their participation and take written consent if agreed. This recruitment process and their participation in the study will not interfere with discharge planning during the study.

Group allocation:

Sealed opaque envelopes contained randomly generated codes for treatment allocations will be given to a member of the clinical team. Once informed consent has been provided, the envelope will be opened randomising participants into two groups: 1) A control group who will conduct conventional sit-to-stand training and 2) An experimental group who will conduct augmented STS training using the feedback system. Twenty participants will be randomly allocated to each group. Participants allocated to either group will be attached with a physical activity monitor (ActivePAL sensor,PAL Technologies Ltd, Glasgow) by the researcher onto the unaffected or dominant side of the thigh. Full instructions will be provided on its use. The monitor is small and lightweight (<15 grams) but capable of detecting and storing information on movement and position (e.g. duration of sitting, standing and the number of STS execution 24 hours aday for 28 days).Data to record from medical notes: Participants' background information (i.e. gender, age, height, weight, reasons for admission and number and type of co-morbidities) will be noted.Pre-assessments:

Participants in both groups will be asked to carry out the following baseline measurements by the researcher: 1)Timed performance of up to five repetitions of the sit to stand movement (FTSTST), if able; 2) Abbreviated Mental Test -4 with a inclusion score of 4 or higher (AMT-4); 3) Tinetti Gait and Balance Assessment (TGBA); 4) Elderly Mobility Scale Test (EMST). These assessments are already being used by the clinical team. Training with the system:The rehabilitation staff will supervise all training sessions as per normal practice. The researcher will provide technical support for all the sessions. The participant will be asked to sit on an adjustable chair with armrests. The height of the chair to be adjusted by the researcher for individual needs. A loose vest with a pouch pocket fitted near the chest region will be worn by the participant. Help will be provided by the researcher if needed. An inertial sensor (Spatial 3/3/3, Phidgets Inc, Calgary, Alberta, Canada) will be placed into the pocket and connected by a USB (Universal Serial Bus) cable to a laptop computer. The participant will then be asked to place both feet on a portable balance plate (BP5046, Bertec Inc, Columbus, OH, USA), which is also attached to the laptop via the USB. The system provides a virtual reality environment that simulates user getting on and off a bus seat. The participant can observe their real-time movement as an avatar on a computerised image (projected on a wall by a projector). Real-time feedback on performance (balance, strength and/or coordination), verbally and visually, will be provided throughout training. The game can be personalised to suit different needs based on the participant's real-time performance. Training should be two to three times a week based on advice on current practice. During the study, the researcher will check with the ward staff that the activity monitor (ActivePAL) is still attached to the participant's thigh and that they are free of skin irritation. The researcher will also change the monitor after seven days so that the skin can be fully inspected and cleaned if necessary. After the study, the monitor will be completely removed by the researcher. The captured anonymised physical activity data will be downloaded to an encrypted folder on a computer and used exclusively for this study. It will then be transferred to a secured computer at the University of Strathclyde for safe storage. Post-assessment: The researcher will carry out a repeat of the baseline measurements at the end of the study.

In addition, the following information will be recorded by the researcher on acceptability and feasibility: 1) Number of sessions attended as a proportion of a total number of the session available; 2)Adverse incidents, type and number; 3) acceptability of the system by a semi-structured interview with the clinical team and participants. The anonymised data will be analysed to address three questions:

1. Is the system feasible to use with older people undergoing inpatient rehabilitation?
2. Is the system feasible to use in a clinical environment?
3. Can the system improve sit-to-stand performance compared to conventional training?
4. Is the system acceptable from the point of view of users (patients and rehabilitation staff)?

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to the geriatric rehabilitation ward at Gartnavel General (Greater Glasgow and Clyde Health Board).
2. Patients with physical impairments that affect their ability to stand up from sitting (sit to stand).
3. Patients that are medically stable.
4. Patients able to give informed consent.
5. Patients able to complete a STS movement with/without the help of a mobility aid or assistance of one other person.
6. Patients able to follow a three-word instruction in English.

Exclusion

1. Patients unable to read feedback on a computer screen with or without the use of visual aids.
2. Patients known to be epileptic/photosensitive or experience blackouts when exposed to certain light patterns or flashing images.
3. Patients with coexisting physical impairments which prevent the practice of sit-to-stand e.g. bilateral amputee or an acute exacerbation of rheumatoid arthritis.
4. Patients not expected to survive during the period of the study
5. Patients with active dermatological problems that may preclude the use of double sided sticky tape.
6. Patients with active medical conditions that may limit prescribed mobility exercise e.g. unstable angina.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-04-18 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
sit to stand ability | 6 weeks
  Five times sit to stand test

SECONDARY OUTCOMES:
Acceptability | 6 weeks
  opinions from users on acceptability of system. This will be gained through semi-structured interviews with participants after completion of the intervention and will be conducted by an independent interviewer. These interviews will be brief (10 mins) and focus on the practicalities of using the system (e.g.length of time to set up) as well as the type of feedback provided. We will aim to interview all the participants (n=20) in the intervention arm.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kerr, Principal Investigator — University of Strathclyde
Locations (1):
- Gartnavel General Hospital, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No